CLINICAL TRIAL: NCT06039033
Title: Merkel Cell Carcinoma Clinical Trials: What Are Prevailing Patient Experiences in Merkel Cell Carcinoma Studies
Brief Title: Exploring Merkel Cell Carcinoma Clinical Trial Engagement Patterns
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 90700326
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Merkel Cell Carcinoma
Keywords: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in medical research usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of Merkel cell carcinoma patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future Merkel cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Able to comprehend the investigational nature of the protocol and provide informed consent
* Diagnosis of Merkel cell carcinoma

Exclusion Criteria:

* No diagnosis of Merkel cell carcinoma confirmed
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Merkel cell carcinoma who are actively considering enrolling in a clinical trial, but have not yet completed enrollment and randomization phases in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a Merkel cell carcinoma clinical research | 3 months
Rate of patients who remain in Merkel cell carcinoma clinical research to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lambert J, Marrel A, D'Angelo SP, Burgess MA, Chmielowski B, Fazio N, Gambichler T, Grob JJ, Lebbe C, Robert C, Russell J, Guzel G, Bharmal M. Patient Experiences with Avelumab in Treatment-Naive Metastatic Merkel Cell Carcinoma: Longitudinal Qualitative Interview Findings from JAVELIN Merkel 200, a Registrational Clinical Trial. Patient. 2020 Aug;13(4):457-467. doi: 10.1007/s40271-020-00428-5. PMID 32472503
- [Background] Kaufman HL, Russell J, Hamid O, Bhatia S, Terheyden P, D'Angelo SP, Shih KC, Lebbe C, Linette GP, Milella M, Brownell I, Lewis KD, Lorch JH, Chin K, Mahnke L, von Heydebreck A, Cuillerot JM, Nghiem P. Avelumab in patients with chemotherapy-refractory metastatic Merkel cell carcinoma: a multicentre, single-group, open-label, phase 2 trial. Lancet Oncol. 2016 Oct;17(10):1374-1385. doi: 10.1016/S1470-2045(16)30364-3. Epub 2016 Sep 1. PMID 27592805
- [Background] Topalian SL, Bhatia S, Amin A, Kudchadkar RR, Sharfman WH, Lebbe C, Delord JP, Dunn LA, Shinohara MM, Kulikauskas R, Chung CH, Martens UM, Ferris RL, Stein JE, Engle EL, Devriese LA, Lao CD, Gu J, Li B, Chen T, Barrows A, Horvath A, Taube JM, Nghiem P. Neoadjuvant Nivolumab for Patients With Resectable Merkel Cell Carcinoma in the CheckMate 358 Trial. J Clin Oncol. 2020 Aug 1;38(22):2476-2487. doi: 10.1200/JCO.20.00201. Epub 2020 Apr 23. PMID 32324435

DOCUMENTS (1):
  • Informed Consent Form (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT06039033/ICF_000.pdf